CLINICAL TRIAL: NCT06934551
Title: Patient Satisfaction & Abutment Teeth Health in Maxillectomy Patients Rehabilitated With Laser CAD CAM & Conventionally Constructed Obturators
Brief Title: Patient Satisfaction & Abutment Teeth Health in Maxillectomy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nehal Abdelrahim Amin Elsherif, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1224
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Maxillary Diseases
MeSH Terms: conditions — Maxillary Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD CA laser polished obturator (Experimental): the intervention obturator is to be made digitally with CAD CAM technology then laser polished
  Interventions: Device: obturator
- conventionally constructed obturator (Active Comparator): the control group will receive conventionally constructed obturator
  Interventions: Device: obturator

INTERVENTIONS:
Device: obturator — conventionally constructed and polished obturator
  Other Names: conventionally constructed obturator

SUMMARY:
randomized controlled trial in maxillectomy patients with two types of obturators with different manufacturing techniques

DETAILED DESCRIPTION:
randomized controlled trial measuring patient satisfaction and abutment teeth health in maxillectomy patients rehabilitated with laser polished CAD CAM obturators versus conventionally constructed obturators

ELIGIBILITY:
Inclusion Criteria

* Patients with hemi maxillectomy
* Sufficient number of natural teeth not less than 5 teeth
* Age between 30 and 60 years
* Intact soft palate

Exclusion Criteria

* Cognitive impairment
* Heavy smokers
* Patients exposed to radiotherapy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 3 months
  will be assessed by 5-point Likert scale capturing various degrees of opinion from strongly disagree, disagree, neutral agree, to strongly agree. data will be collected and sent to statistician for the analysis required in mean difference and standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No